CLINICAL TRIAL: NCT04857073
Title: Daily Versus Every Other Day Glucose Monitoring in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Kristina Feldman, Maternal Fetal Medicine Fellow, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 20-01914
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Gestational Diabetes
Keywords: glucose monitoring
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two arms
  1. daily, 4 times a day glucose monitoring (fasting, 2 hours post prandial x 3)
  2. every other day, 4 times daily glucose monitoring (fasting, 2 hours post prandial x 3)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - glucose check every day (Active Comparator): Patients will be instructed to check their glucose 4 times a day, every day. This is currently the standard of care.
  Interventions: Other: Glucose Monitoring
- Experimental group - glucose check every other day (Experimental): Patients will be instructed to check their glucose every other day, 4 times glucose monitoring
  Interventions: Other: Glucose Monitoring

INTERVENTIONS:
Other: Glucose Monitoring — Glucose monitoring consists of finger stick fasting and 2 hours post prandial
  Other Names: Fingerstick

SUMMARY:
Gestational diabetes mellitus (GDM) occurs secondary to carbohydrate intolerance in pregnancy. Screening of GDM occurs between 24 to 28 weeks gestation by a screening 1-hour 50g glucose challenge test and confirmed with a 100g 3-hour fasting glucose tolerance test. Once patients are diagnosed with GDM, they are instructed to check their fingerstick blood glucose four times daily, every day. There is insufficient evidence to determine the ideal frequency and timing of glucose monitoring in patients diagnosed with GDM and no absolute guidelines put in place by the American College of Obstetricians and Gynecologists (ACOG). The study team aims to confirm non inferiority on the patient population on the effects of daily (4x daily) versus every other day (4x daily) glucose monitoring in all patients diagnosed with GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) occurs secondary to carbohydrate intolerance in pregnancy. Screening of GDM occurs between 24 to 28 weeks gestation by a screening 1-hour 50g glucose challenge test and confirmed with a 100g 3-hour fasting glucose tolerance test. In the study team's practice, once a patient is diagnosed with GDM, they are enrolled in the Diabetes in Pregnancy program, undergo nutritional education, diabetes education and have their care overseen by a Maternal-Fetal Medicine specialist. They are instructed to check their fingerstick blood glucose four times daily, every day. There is insufficient evidence to determine the ideal frequency and timing of glucose monitoring in patients diagnosed with GDM and no absolute guidelines put in place by the American College of Obstetricians and Gynecologists. In 2017, a randomized control trial was performed by Menedez-Figeroa et al, showing non inferiority in patients diagnosed with GDM who were instructed to perform every other day (4 time daily) glucose monitoring versus daily (4 times daily) glucose monitoring with their primary outcome being a 5% change in birthweight between groups at delivery. The study team aims to confirm non inferiority on the patient population on the effects of daily (4x daily) versus every other day (4x daily) glucose monitoring in all patients diagnosed with GDM with the primary outcome being a 0% difference in birth weight. The study team will be enrolling approximately 300 patients. If a patient is enrolled in the study, there will be no excursion from normally scheduled visits (including follow ups), medications regimens, or procedure (including ultrasounds). They will remain in the Diabetes in Pregnancy program throughout their pregnancy. Participants will be enrolled at the first visit with the high risk doctor, and they will be asked to perform standard (4x daily) fingerstick monitoring, or every other day fingerstick monitoring (4x daily, every other day). Data collected from the patient (including labs, and fingerstick glucose values) will not be exclusively for research purposes, and will be collected as a routine part of the patients care

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies in women 18 years or older
* Diagnosis of GDM between 24 to 28 weeks gestation

Exclusion Criteria:

* Preexisting diabetes mellitus or GDM diagnosed prior to 24 weeks by early GDM screening (including patients currently on insulin or any oral hypoglycemic agent)
* Diagnosis of GDM based on fingerstick paneling
* Women who are on chronic steroid therapy
* Multifetal gestation
* Patients with GTT fasting value >100 (which would indicate a diagnosis of pre-diabetes according to the American Diabetes Association)
* Patients who exhibited poor compliance after the first two weeks of glucose monitoring (which is defined as less than 20% of expected values recorded during the 2 week period of initial testing)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Birth weight | Day 1 - day of delivery
  Fetal weight at time of delivery (grams).

SECONDARY OUTCOMES:
APGAR score | Day 1 - day of delivery
  APGAR measures the baby's color, heart rate, reflexes, muscle tone, and respiratory effort and total score from 1 to 10, with higher score indicating better health outcomes
Cord blood pH level | Day 1 - day of delivery
Number of NICU admission | Day 1 - day of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Feldman, DO, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Perinatal Associates, New York, New York, United States

REFERENCES:
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Derived] Feldman KM, Coughlin A, Feliciano J, Stoffels G, Wang KZ, Strauss TS, Grubman O, Al-Ibraheemi Z, Cole D, Ashmead G, Hussain F, Shchur SS, Lee D, Brustman L. Neonatal Birth Weight With Daily Compared With Every-Other-Day Glucose Monitoring in Gestational Diabetes Mellitus: A Randomized Controlled Trial. Obstet Gynecol. 2024 Nov 1;144(5):707-714. doi: 10.1097/AOG.0000000000005528. Epub 2024 Feb 8. PMID 38330409